CLINICAL TRIAL: NCT02086825
Title: A Randomized Comparison of Rifaximin Versus Lactulose in Hospitalized Cirrhotic Patients With Renal Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-00665
Record Dates: First submitted 2014-02-11; First posted 2014-03-13 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental)
  Interventions: Drug: Rifaximin
- Lactulose (Experimental)
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Rifaximin — (Xifaxin®, Salix Pharmaceuticals) 550mg tablet twice daily.
  Other Names: Xifaxin
  Arms: Rifaximin
Drug: Lactulose — 20g dose titrated
  Arms: Lactulose

SUMMARY:
The aim of the current study is to determine whether rifaximin or lactulose is more effective in preventing the development of severe hepatic encephalopathy in hospitalized patients with cirrhosis and new onset kidney failure.

Subjects will be randomly assigned to one of two treatment groups:

Group A: Lactulose 20g dose titrated to 2-3 soft-formed bowel movements per day Group B: Rifaximin 550mg tablet twice daily.

Subjects will be followed daily for two weeks or until hospital discharge. Treatment success is defined as prevention of grade 3 or 4 HE during hospitalization.

DETAILED DESCRIPTION:
Hepatic Encephalopathy (HE) is a reversible neuropsychiatric syndrome that develops in patients with cirrhosis due to the accumulation of a variety of toxic substances that are produced from bacteria in the gastrointestinal tract. It is characterized by slowing of function of the brain function and ranges in severity from mild cognitive impairment (grade 1), presence of a shaking tremor called asterixis (grade 2), lethargy but arousable state (grade 3), and coma (grade 4). Decreased kidney function exacerbates the condition, and hospitalized patients with cirrhosis with new onset kidney failure are at risk for the development of severe HE.

Possible treatments for HE include lactulose and antibiotics. Lactulose reduces the production of many of the toxins by the bacteria, and antibiotics work by reducing the number of bacteria in the gastrointestinal tract. Rifaximin is an antibiotic that is an antibiotic that is not absorbed, possesses a wide antibacterial spectrum, and was approved by the Food and Drug Administration in 3/2010 for prevention of relapse for patients with recurrent severe hepatic encephalopathy. The aim of the current study is to determine whether rifaximin or lactulose is more effective in preventing the development of severe hepatic encephalopathy in hospitalized patients with cirrhosis and new onset kidney failure.

To determine whether rifaximin or lactulose is more effective in preventing severe HE, seventy consecutive hospitalized patients with cirrhosis and new onset kidney failure will be recruited. New onset kidney failure will defined as a progressive and sustained increase in serum creatinine >0.5mg/dl from baseline to a value of 2.0mg/dl or greater within 3 days. Subjects will be randomly assigned to one of two treatment groups:

Group A: Lactulose 20g dose titrated to 2-3 soft-formed bowel movements per day Group B: Rifaximin 550mg tablet twice daily. Subjects will be followed daily for two weeks or until hospital discharge. Severity of hepatic encephalopathy will be graded by physical examination, review of hospital chart, and performance of standard paper and pencil tests that evaluates the ability to concentrate. In addition, approximately one tablespoon will be drawn twice a week at every 3 to 4 day for ammonia level and other toxins. A sample of breath will also be collected by having the subjects breathe into a collection bag to measure substances that determine whether there are bacteria present in the small intestine. Treatment success is defined as prevention of grade 3 or 4 HE during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Cirrhosis of the liver based on biopsy or clinical and radiographic criteria
3. Ability to provide informed consent (Grade 0 to 1 HE)
4. Acute renal failure (increase in baseline creatinine of 0.5mg/dL to a value of >2.0 mg/dL within 3 days).
5. Absence of improvement in renal function after adequate fluid resuscitation using either normal saline or blood products (25% salt poor albumin, fresh frozen plasma, or packed red blood cells)

Exclusion Criteria:

1. Previous history of sensitivity/allergy to lactulose or rifaximin or rifampin
2. Pregnancy
3. Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Development of Progressive Hepatic Encephalopathy to Stage 3 or 4 in patients with progressive renal failure | 90 days (including follow-ups)
  The primary outcome for this study is the development of progressive hepatic encephalopathy to stage 3 or 4 in patients with progressive renal failure. For the purpose of this study, acute renal failure is defined as a progressive and sustained increase in serum creatinine >0.5mg/dl from baseline to a value of 2.0mg/dl, irrespective of etiology in 3 days. Renal failure is progressive and sustained if there is no improvement after volume resuscitation with 1.5 L of normal saline or equivalent colloid infusion (serum albumin or blood product transfusion).

SECONDARY OUTCOMES:
In-hospital mortality | Patient's hospital stay up to 14 days
Hospital Length of Stay | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- New York University Langone Medical Center, New York, New York, United States